CLINICAL TRIAL: NCT03312660
Title: Effect of a Kefir Beverage on Immunity and Lipid Profile: An Exploratory Cluster Randomized Controlled Trial
Brief Title: Effect of a Kefir Beverage on Immunity and Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Maria del Mar Calvo Malvar, Principal Investigator, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INNTER BIOFUNCIOGAL 2015
Record Dates: First submitted 2017-10-04; First posted 2017-10-18 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Prebiotics
Keywords: Prebiotics; kefir
MeSH Terms: interventions — Cultured Milk Products; Dairy Products

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both groups will receive fermented dairy products with similar color, flavor and nutritional composition, except the prebiotic components, which will only be administered to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic group. (Experimental): Group of 22 families consuming a fermented dairy product with prebiotic components, once a day for 4 months.
  Interventions: Dietary Supplement: Prebiotic group
- Placebo group (Placebo Comparator): Group of 22 families consuming a dairy product with similar characteristics regarding color, flavor and nutritional composition, not containing the prebiotic components, once a day for 4 months.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Prebiotic group — Fermented dairy product with galacto-oligosaccharides (GOS), kefiran and other metabolites resulting from the fermentation with kefir granules.
  Other Names: Fermented dairy product with kefir granules
  Arms: Prebiotic group.
Dietary Supplement: Placebo group — Beverage with color, flavor and nutritional composition similar to the fermented dairy product but not containing the prebiotic components.
  Other Names: Dairy product without prebiotic components
  Arms: Placebo group

SUMMARY:
This is an exploratory cluster randomized controlled trial to evaluate the effect of a kefir beverage, enriched with prebiotics components, on immunity, lipid profile and adiposity in a population-based study, using the family as the intervention unit.

DETAILED DESCRIPTION:
The gastrointestinal tract is populated by a collection of microorganisms, primarily bacteria, that interact with intestinal host cells. In the past two decades, several studies have demonstrated the effects of the intestinal microbiota on host physiological, metabolic and immunological processes and have revealed that the microbiota is fundamental to host body function. There is currently a growing interest in manipulating the intestinal microbiota to enhance the effects on health and welfare of the intestine. In this regard, since its introduction, the concept of prebiotics has stimulated both scientific and industrial interest. A dietary prebiotic is a selectively fermented ingredient that results in specific changes, in the composition and/or activity of the gastrointestinal microbiota, thus conferring benefits upon host health. To date, the prebiotics most widely evaluated in human clinical trials are inulin-type fructans (inulin, fructo-oligosaccharides, oligofructose) and galacto-oligosaccharides (GOS).

The investigators goal is to conduct a human clinical trial to evaluate the impacts of a functional-prebiotic beverage on immunity and metabolic profile.

This study will be performed on a family-oriented basis. 44 families/clusters (~ 150 children and adults, older than 3 years) will be selected to participate in the study and will be randomized into intervention group (n=22 families) and control (n=22 families) groups.

Weight, body mass index (BMI), waist circumference (WC), nutrient intake from food frequency questionnaire, physical activity, blood pressure, allergic sensitization, metabolic function (fasting blood glucose, HbA1c, insulin resistance and lipid profile), general lymphocyte overview (B-cells, T-cells and NK-cells) and sub-populations of T-helper cells (Th1, Th2, Th17 and T-regulatory), inflammation markers (C-reactive protein, interleukin-6 and tumor necrosis factor-alpha) will be measured at baseline and after 4 months.

Mixed effect models analysis will be performed to assess changes in the cardiometabolic and immune parameters.

ELIGIBILITY:
Inclusion Criteria:

1. For the index subject:

   * Female or male.
   * 18 years and older.
   * Living in a family unit with two or more people.
2. For the other family members:

   * Female or male.
   * Age between 3 to 85 years.
3. At family level: at least two members will meet inclusion criteria but no exclusion criterion

Exclusion Criteria for the index subject and the other family members:

* Alcoholism
* Pregnant
* Major cardiovascular disease
* Dementia
* Major autoimmune diseases
* Diseases or treatments that seriously affect the immune status
* Neoplasia
* Terminal disease

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Th17 cell counts in peripheral blood | 4 months
  Flow cytometry analysis on peripheral blood
Change from baseline in CD4 positive regulatory T cell counts in peripheral blood | 4 months
  Flow cytometry analysis on peripheral blood
Change from baseline in Th1 cell counts in peripheral blood | 4 months
  Flow cytometry analysis on peripheral blood
Change from baseline in Th2 cell counts in peripheral blood | 4 months
  Flow cytometry analysis on peripheral blood

SECONDARY OUTCOMES:
Change from baseline in total cholesterol | 4 months
  Enzymatic method using standard kits on an Advia 2400 Clinical Chemistry System (Siemens Healthcare Diagnostics)
Change from baseline in HDL cholesterol | 4 months
  Enzymatic method using standard kits on an Advia 2400 Clinical Chemistry System (Siemens Healthcare Diagnostics)
Change from baseline in LDL cholesterol | 4 months
  Estimated using the Friedewald formula. Enzymatic method when triglycerides > 400 mg/dl.
Change from baseline in triglycerides | 4 months
  Enzymatic method using standard kits on an Advia 2400 Clinical Chemistry System (Siemens Healthcare Diagnostics)
Change from baseline in allergic sensitization measured through a battery of 11 skin prick test to common allergens | 4 months
  Cases with at least one positive test will be considered to have allergic sensitization.
Change from baseline in B lymphocytes in peripheral blood | 4 months
  Flow cytometry analysis on peripheral blood
Change from baseline in T lymphocytes in peripheral blood | 4 months
  Flow cytometry analysis on peripheral blood
Change from baseline in Natural Killer (NK) lymphocytes in peripheral blood | 4 months
  Flow cytometry analysis on peripheral blood
Change from baseline in C-reactive protein | 4 months
  Immunometric chemoluminiscence method employing an Immulite 2000 Immunoassay System
Change from baseline in interleukin-6 | 4 months
  Immunometric chemoluminiscence method employing an Immulite 2000 Immunoassay System
Change from baseline in tumor necrosis factor-alpha | 4 months
  Immunometric chemoluminiscence method employing an Immulite 1000 Immunoassay System
Change from baseline in glucose | 4 months
  Enzymatic method using standard kits on an Advia 2400 Clinical Chemistry System (Siemens Healthcare Diagnostics)
Change from baseline in HbA1c | 4 months
  High resolution liquid chromatography using a Menarini Diagnostics HA-8160 Analyzer;
Change from baseline in insulin | 4 months
  Immunometric chemoluminiscence method employing an Immulite 2000 Immunoassay System
Change from baseline in body mass index (BMI) | 4 months
  BMI will be calculated as body weight (kg) divided by height (m) squared. The BMI of subjects under 18 years of age will be standardised using World Health Organization (WHO) reference data.
Change from baseline in waist circumference | 4 months
  Waist circumference will be measured at the narrowest point between the bottom rib and the top of the iliac crest.
Change from baseline in hip circumference | 4 months
  Hip circumference will be measured at the point of greatest prominence of the gluteal muscles.
Change from baseline in stool frequency | 4 months
  Evaluated through a questionnaire.
Change from baseline in stool consistency (Bristol Stool Form Scale score) | 4 months
  Bristol Stool Form Scale (BSFS) is for classifying the form of stool into 7 categories scored from 1 to 7; (1) Separate hard lumps like nuts (difficult to pass); (2) Sausage-shaped but lumpy; (3) Like a sausage but with cracks on its surface; (4) Like a sausage or snake, smooth and soft; (5) Soft blobs with clear-cut edges (passed easily); (6) Fluffy pieces with ragged edges, a mushy stool; (7) Watery, no solid pieces, entirely liquid. Subjects choose one of the BSFS scores which has a nearest analog form with their stools at every defecation.
  Types 1 and 2 are considered to be abnormally hard stools, while Types 6 and 7 are considered abnormally liquid stools. Types 3, 4 and 5 are generally considered to be the most normal stool forms.
Change from baseline in food intake over the last 4 weeks | 4 months
  Assessed using a semi-quantitative food frequency questionnaire (FFQ) which include 93 foods and drinks habitually consumed in Spain.

CONTACTS AND LOCATIONS:
Overall Officials: Mar Calvo-Malvar, PhD, Study Chair — Clinic University Hospital of Santiago, Santiago de Compostela, Spain.
Locations (1):
- A Estrada Primary Care Centre, A Estrada, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No